CLINICAL TRIAL: NCT00371696
Title: Pilot Study of the Feasibility of n-of-1 Trials: the Individualisation of Treatments for Osteoarthritis
Brief Title: Feasibility of n-of-1 Trials - a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bristol (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: SMD LREC 108/01
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2003-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac; Acetaminophen

INTERVENTIONS:
Drug: diclofenac
Drug: paracetamol
Device: heat retaining knee support
Device: standard knee support

SUMMARY:
The aim of this study was to provide essential pilot data on the feasibility of conducting n-of-1 trials within secondary care within the UK, notably to: test the process of recruitment and design aspects of such trials; assess the acceptability of this research method to patients, explore the experiences of patients involved; determine the most appropriate treatment for individual patients.

DETAILED DESCRIPTION:
Whilst the large scale randomised controlled trial (RCT) remains the scientific "gold standard" for evaluating therapies in clinical medicine, the assumption made, that the treatment effect demonstrated is generalisable and applicable to all patients, is unlikely to be true. There will inevitably be some patients who benefit from a particular treatment more than others. N-of-1 trials are a means of conducting RCTs in individual patients with the added opportunity to use patient generated outcome measures. Patients act as their own control and receive all treatments under comparison, more than once, in a random sequence. While n-of-1 trial methodology is reasonably well specified they remain under-exploited and little is known about the process aspects of conducting such trials or the experiences and views of those who participate in them. The time commitment by patients and health professionals is not inconsiderable and there may well be particular problems with recruitment and drop out. N-of-1 trials rely on co-operation between individual clinicians and patients, however, no work has been undertaken to explore the ways in which patient-practitioner relationships and their experiences and views influence the progress and outcome of n-of-1 trials.

Patients with confirmed osteoarthritis (OA) of the knee, selected for a mix of gender, age, weight, will be recruited to the n-of-1 trials to compare either, an NSAID (diclofenac) with simple analgesic (paracetamol) or a standard knee support with a heat retaining support. Patients will undergo a (1 hour) semi-structured interview before the trial commences and once the trial is completed or terminated. Patients treated with supports/drugs will receive each treatment for a period of one/two weeks respectively, for 3 cycles (order determined at random). Patients will complete daily diaries including standard patient questionnaires and a patient generated outcome measure. Qualitative interviews and observational methods will be employed to study practitioner/ patient relationships; decision to participate; expectations and experience; appropriateness and acceptability of research design and measures. Patients declining to take part will be approached to explore reasons for not participating.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending clinics in the North Bristol Health Care Trust, with confirmed OA of the knee (Kellgren-Lawrence radiographic score of 2-4 within the previous 12 months) and use-related pain.

Exclusion Criteria:

* Patients who had received corticosteroid injections or operations on their knee in the previous six months were excluded. Those with known contraindications to paracetamol or any NSAID, and those taking steroids, warfarin or aspirin for another medical condition were excluded from the drug trials.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2001-12; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dieppe, Study Director — MRC Health Services Research Collaboration
Locations (1):
- Southmead Hospital, Bristol, United Kingdom